CLINICAL TRIAL: NCT04937296
Title: Effects of a Home-based Physical Activity Programme on Blood Biomarkers and Health-related Quality of Life Indices in Saudi Arabian Type-2 Diabetes Mellitus Patients: a Pilot Randomised Controlled Trial
Brief Title: Effects of Home-based Physical Activity in Saudi Arabian Type-2 Diabetes Mellitus Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Sinclair (Other)
Collaborators: University of Hertfordshire (Other); University of Jazan (Other Government)
Responsible Party: Sponsor-Investigator, Jonathan Sinclair, Research professor, University of Central Lancashire
Organization: University of Central Lancashire (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Home based physical activity
Record Dates: First submitted 2021-06-14; First posted 2021-06-24 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Placebo Comparator)
  Interventions: Other: Usual care
- Physical activity (Experimental)
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — Participants will be asked to perform resistance exercises 3-times a week on alternating days for 12 weeks. Exercises will be performed with a TheraBand and will include the squat, lunge, press-up, cross body reach, reverse fly, lateral raise, biceps curl, triceps extension, frontal raise and bridge. In addition to the resistance exercises, the participants will perform aerobic exercise. They will be asked to download a specific exercise app to record the number of steps on day 1 of the intervention and participants who do not possess the required phone technology will be provided with a pedometer. They then will be asked to add 2000 steps on to their daily steps; this amount will then become their daily step goal. Once they have reached this goal on 4 out of 5 days, they will be asked to increase their new step step goal by an extra 500 per day.
  Arms: Physical activity
Other: Usual care — Usual care.
  Arms: Usual care

SUMMARY:
The World Health Organization ranks Saudi Arabia as having the 7th highest rate of type-2 diabetes in the world. This therefore makes diabetes the most challenging health problem facing Saudi Arabia. Importantly, physical activity has been shown to improve disease symptoms and overall health in patients with type-2 diabetes. However, findings relating to the prevalence of physical inactivity in the Saudi population confirm that a sedentary lifestyle is on the rise, within physical inactivity levels in adults being 80.5%. Therefore, interventions aimed at reducing physical inactivity using bespoke modalities pertinent to Saudi Arabia are clearly warranted.

The purpose of this research project is to undertake a feasibility randomised control trial, examining the effects of a 12-week home-based physical activity programme on HbA1c, blood lipids, fasting glucose and other indices of health-related quality of life in Saudi Arabian adults with type-2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Clinically established diagnosis of type-2 diabetes for at least 12 months
* Previously sedentary
* Knowledgeable about hypoglycemia
* Aged over 18 years
* Capacity to give informed consent.

Exclusion Criteria:

* Cognitive impairment precluding consent or participation
* Pregnancy
* Additional medical conditions that prevent safe physical activity (e.g. severe arthritis or advanced heart failure)
* Enrolment in any other clinical trial designed to influence type-2 diabetes symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
HBA1c (Glycated hemoglobin) | Baseline
  Glycated hemoglobin is a form of hemoglobin that is chemically linked to a sugar. This parameter will be obtained via a venous blood sample.
HBA1c (Glycated hemoglobin) | 12 weeks
  Glycated hemoglobin is a form of hemoglobin that is chemically linked to a sugar. This parameter will be obtained via a venous blood sample.
HBA1c (Glycated hemoglobin) | 24 weeks
  Glycated hemoglobin is a form of hemoglobin that is chemically linked to a sugar. This parameter will be obtained via a venous blood sample.

SECONDARY OUTCOMES:
WHO Well-Being Index (WHO-5) | Baseline
  The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing. A score of 0 represents the worst imaginable well-being and 100 represents the best imaginable well-being.
WHO Well-Being Index (WHO-5) | 12 weeks
  The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing. A score of 0 represents the worst imaginable well-being and 100 represents the best imaginable well-being.
WHO Well-Being Index (WHO-5) | 24 weeks
  The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing. A score of 0 represents the worst imaginable well-being and 100 represents the best imaginable well-being.
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  The Patient Health Questionnaire-9 (PHQ-9) is the depression module, which has nine questions ranging from "0" (not at all) to "3" (nearly every day). The scoring is interpreted as 0-4 no depression symptoms, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe depression symptoms.
Patient Health Questionnaire-9 (PHQ-9) | 12 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is the depression module, which has nine questions ranging from "0" (not at all) to "3" (nearly every day). The scoring is interpreted as 0-4 no depression symptoms, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe depression symptoms.
Patient Health Questionnaire-9 (PHQ-9) | 24 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is the depression module, which has nine questions ranging from "0" (not at all) to "3" (nearly every day). The scoring is interpreted as 0-4 no depression symptoms, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe depression symptoms.
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality. The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Pittsburgh Sleep Quality Index (PSQI) | 12 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality. The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Pittsburgh Sleep Quality Index (PSQI) | 24 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality. The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Physical fitness | Baseline
  Physical fitness will be examined via the Chester Step test.
Physical fitness | 12 weeks
  Physical fitness will be examined via the Chester Step test.
Physical fitness | 24 weeks
  Physical fitness will be examined via the Chester Step test.
Fasting glucose | Baseline
  Fasting glucose levels will be examined via a venous blood sample.
Fasting glucose | 12 weeks
  Fasting glucose levels will be examined via a venous blood sample.
Fasting glucose | 24 weeks
  Fasting glucose levels will be examined via a venous blood sample.
Systolic blood pressure | Baseline
  Systolic blood pressure using blood pressure monitor with blood pressure cuff on the arm.
Systolic blood pressure | 12 weeks
  Systolic blood pressure using blood pressure monitor with blood pressure cuff on the arm.
Systolic blood pressure | 24 weeks
  Systolic blood pressure using blood pressure monitor with blood pressure cuff on the arm.
Diastolic blood pressure | Baseline
  Diastolic blood pressure using blood pressure monitor with blood pressure cuff on the arm.
Diastolic blood pressure | 12 weeks
  Diastolic blood pressure using blood pressure monitor with blood pressure cuff on the arm.
Diastolic blood pressure | 24 weeks
  Diastolic blood pressure using blood pressure monitor with blood pressure cuff on the arm.
Lipid profile | Baseline
  A full lipid profile will be undertaken this involves Low-density lipoprotein (LDL), High-density lipoprotein (HDL), Triglycerides and Total cholesterol levels. This will be examined via a venous blood sample.
Lipid profile | 12 weeks
  A full lipid profile will be undertaken this involves Low-density lipoprotein (LDL), High-density lipoprotein (HDL), Triglycerides and Total cholesterol levels. This will be examined via a venous blood sample.
Lipid profile | 24 weeks
  A full lipid profile will be undertaken this involves Low-density lipoprotein (LDL), High-density lipoprotein (HDL), Triglycerides and Total cholesterol levels. This will be examined via a venous blood sample.
Body mass | Baseline
  Body mass in kg measured via an electric scale.
Body mass | 12 weeks
  Body mass in kg measured via an electric scale.
Body mass | 24 weeks
  Body mass in kg measured via an electric scale.
Body mass index | Baseline
  Body mass index will be quantified using the standard body mass index equation using measures of body mass and stature.
Body mass index | 12 weeks
  Body mass index will be quantified using the standard body mass index equation using measures of body mass and stature.
Body mass index | 24 weeks
  Body mass index will be quantified using the standard body mass index equation using measures of body mass and stature.
Triglyceride-glucose index | Baseline
  The triglyceride-glucose index will be calculated using a logarithm of the fasting triglyceride and glucose indices.
Triglyceride-glucose index | 12 weeks
  The triglyceride-glucose index will be calculated using a logarithm of the fasting triglyceride and glucose indices.
Triglyceride-glucose index | 24 weeks
  The triglyceride-glucose index will be calculated using a logarithm of the fasting triglyceride and glucose indices.

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan Diabetes Centre, Jizan, Saudi Arabia